CLINICAL TRIAL: NCT00667290
Title: Exercise for Elderly Peripheral Revascularized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Andrew W. Gardner, PhD, CMRI Hobbs-Recknagel Professor, University of Oklahoma Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0098; R01AG016685 (NIH)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
Keywords: functional ability; gait; musculoskeletal disorder therapy; peripheral blood vessel disorder
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Treadmill exercise
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Treadmill exercise — Graded treadmill walking 3 times per week for 3 months
  Arms: 1

SUMMARY:
The purpose of this study is (1) to determine whether a 3-month exercise rehabilitation program will improve claudication distances, free-living daily physical activity, and health-related quality of life of older, revascularized patients with peripheral arterial disease, and (2) to determine whether the primary mechanisms by which exercise rehabilitation affects the above functional outcomes are through alterations in walking efficiency, peripheral circulation, and cardiopulmonary function.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) patients with critical limb-threatening ischemia have improved peripheral circulation following infrainguinal revascularization. Despite this hemodynamic benefit, little change in functional status occurs, and many patients have residual ambulatory dysfunction. The lack of functional improvement in revascularized patients may be due to extreme physical deconditioning secondary to their pre-existing critical limb-threatening ischemia. Therefore, we hypothesize that a program of aerobic exercise training is necessary to optimize ambulation, free-living daily physical activity, and health-related quality of life through the mechanisms of improved walking economy, peripheral circulation, and cardiopulmonary function.

This is a prospective, randomized controlled clinical trial comparing an exercise group undergoing a program of graded treadmill walking, and a non-exercise control group. Eighty PAD patients will be randomized into either the exercise group (N = 40) or the non-exercise control group (N = 40) following successful lower extremity arterial bypass or angioplasty. The 3-month exercise program will consist of graded treadmill walking 3 times per week with progressive increments in exercise duration from 15 to 40 minutes, and progressive increments in exercise intensity from 50 to 80% of exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* lower extremity arterial bypass at least 3 months prior to screening
* infrainguinal percutaneous transluminal angioplasty (PTLA) at least 2 weeks prior to screening

Exclusion Criteria:

* persistent rest pain due to (peripheral artery disease (PAD) (Fontaine Stage III for PAD),
* persistent tissue loss due to PAOD (Fontaine Stage IV for PAD),
* medical conditions that are contraindicative for exercise according to the American College of Sports Medicine (e.g., acute myocardial infarction, unstable angina, etc.)
* cognitive dysfunction (mini-mental state examination score of less than 24)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2000-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in the walking distance to onset of leg pain, and the change in walking distance to maximal leg pain

SECONDARY OUTCOMES:
Changes in walking efficiency, calf muscle circulation, and cardiopulmonary function.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W. Gardner, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- General Clinical Research Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Gardner AW, Katzel LI, Sorkin JD, Bradham DD, Hochberg MC, Flinn WR, Goldberg AP. Exercise rehabilitation improves functional outcomes and peripheral circulation in patients with intermittent claudication: a randomized controlled trial. J Am Geriatr Soc. 2001 Jun;49(6):755-62. doi: 10.1046/j.1532-5415.2001.49152.x. PMID 11454114
- [Background] Gardner AW, Katzel LI, Sorkin JD, Goldberg AP. Effects of long-term exercise rehabilitation on claudication distances in patients with peripheral arterial disease: a randomized controlled trial. J Cardiopulm Rehabil. 2002 May-Jun;22(3):192-8. doi: 10.1097/00008483-200205000-00011. PMID 12042688
- [Background] Gardner AW, Killewich LA, Montgomery PS, Katzel LI. Response to exercise rehabilitation in smoking and nonsmoking patients with intermittent claudication. J Vasc Surg. 2004 Mar;39(3):531-8. doi: 10.1016/j.jvs.2003.08.037. PMID 14981444
- [Background] Gardner AW, Montgomery PS, Flinn WR, Katzel LI. The effect of exercise intensity on the response to exercise rehabilitation in patients with intermittent claudication. J Vasc Surg. 2005 Oct;42(4):702-9. doi: 10.1016/j.jvs.2005.05.049. PMID 16242558